CLINICAL TRIAL: NCT04088890
Title: Phase I/Ib Clinical Trial of Autologous CD22 Chimeric Antigen Receptor (CAR) T Cells in Adults With Recurrent or Refractory B Cell Malignancies
Brief Title: Autologous CD22 CAR T Cells in Adults w/ Recurrent or Refractory B Cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Leukemia and Lymphoma Society (Other); American Society of Hematology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-50836; NCI-2019-06810 (Registry Identifier: NCI-CTRP); 5K08CA248968-05 (NIH)
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: B-ALL; B-cell Non Hodgkin Lymphoma; DLBCL; Follicular Lymphoma Grade 3B
Keywords: CD22; CAR T cells
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- R/R ALL (Experimental): Relapsed/refractory ALL
  Lymphodepletion prior to CD22 CAR T cell infusion (Day 0) will occur as follows:
  * Fludarabine 30 mg/m2 per day IV for days 5, 4, 3
  * Cyclophosphamide 500 mg/m2 per day IV for days 5, 4, 3
  Autologous CD22 CAR T cells will be administered intravenously at Dose1: 3 x 10^5cells/kg (± 20%) 10
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: CD22 CAR
- R/R aggressive B-cell NHL (Experimental): Relapsed/refractory aggressive B-cell non-Hodgkin lymphoma.
  Lymphodepletion prior to CD22 CAR T cell infusion (Day 0) will occur as follows:
  * Fludarabine 30 mg/m2 per day IV for days 5, 4, 3
  * Cyclophosphamide 500 mg/m2 per day IV for days 5, 4, 3
  Autologous CD22-CAR T cells will be administered in 3 escalating doses (Dose Level 1, 2, and 3) to determine MTD/RP2D.
  Dose1: 1 x 10^6 cells/kg (± 20%) Dose2: 3 x 10^6 cells/kg (± 20%) Dose3: 1 x 10^7 cells/kg (± 20%)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: CD22 CAR

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2
Drug: Cyclophosphamide — Cyclophosphamide 500 mg/m2
Drug: CD22 CAR — Autologous T cells transduced with lentiviral vector (CD22.BB.Z) Chimeric Antigen Receptor (CD22 CAR). Autologous CD22 CAR T cells will be administered intravenously at Dose Level 1 in subjects with ALL. Autologous CD22-CAR T cells will be administered in 3 escalating doses (Dose Level 1, 2, and 3) in subjects with aggressive B-cell NHL to determine MTD/RP2D

SUMMARY:
The primary purpose of this study is to test whether CD22-CAR T cells can be successfully made from immune cells collected from adults with relapsed/refractory B-cell malignancies (leukemia and lymphoma).

DETAILED DESCRIPTION:
Primary Objective:

* Determine the feasibility of manufacturing CD22 CAR T cells using the Miltenyi CliniMACS Prodigy® system for administration to adults with relapsed/refractory CD22 expressing B-cell ALL or relapsed/refractory aggressive B-cell non hodgkins lymphoma (NHL).
* Establish the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of CD22 CAR T cells in adults with relapsed/refractory aggressive B-cell NHL.
* Determine the safety of an established dose of CD22-CAR T cells in adults with relapsed/refractory CD22 expressing B-cell ALL and the safety of the MTD/RP2D of CD22-CAR T cells in adults with relapsed/refractory aggressive B-cell NHL.

Secondary Objective:

- Assess the clinical activity of CD22-CAR T cells in adults with R/R CD22 expressing B-cell ALL and R/R aggressive B-cell NHL, including overall survival (OS) and progressive free survival (PFS).

ELIGIBILITY:
Inclusion criteria.

1. Disease Status

   1. Disease Status of ALL

      * Must have chemotherapy refractory disease defined as progression or stable disease after two lines of therapies, or relapsed disease after achieving CR.
      * Subjects with persistent or relapsed minimal residual disease (MRD) (by flow cytometry, PCR, FISH, or next generation sequencing) require verification of MRD on two occasions at least 2 weeks apart.
      * Subjects with Philadelphia Chromosome positive acute lymphoblastic leukemia (Ph+ALL) are eligible if they progressed, had stable disease or relapsed after two lines of therapy, including tyrosine kinase inhibitors (TKIs).
      * Subjects with recurrence of isolated CNS relapse after achieving complete remission (CR) are eligible.
   2. Disease Status of aggressive B-cell NHL •Histologically confirmed aggressive B cell NHL including the following types defined by WHO 2008: oDLBCL not otherwise specified; T cell/histiocyte rich large B cell lymphoma; DLBCL associated with chronic inflammation; Epstein Barr virus (EBV)+ DLBCL of the elderly; OR oprimary mediastinal (thymic) large B cell lymphoma; OR otransformation of follicular lymphoma, marginal zone lymphoma or chronic lymphocytic leukemia/small lymphocytic lymphoma to DLBCL; OR oFollicular Lymphoma Grade 3B •Subjects with DLBCL, Follicular Lymphoma Grade 3B -or-

   Subjects with transformed FL, MZL, or CLL/SLL who HAVE NOT received chemotherapy prior to transformation:

   oMust have received an anthracycline regimen and an anti CD20 monoclonal antibody (unless documented CD20-negative) and be refractory or relapsed after second line of DLBCL treatment. Subjects with a partial response to second line therapy must be ineligible for autologous transplant.

   •Subjects with transformed FL, MZL, or CLL/SLL who HAVE received anthracycline-containing chemotherapy prior to transformation: oMust have progressed, had SD or recurred with transformed disease after initial treatment for DLBCL.
2. Measureable Disease

   * Subjects with ALL: must have evaluable or measurable disease (MRD positive by flow cytometry, NGS, or PCR is acceptable).
   * Subjects with aggressive B-cell NHL: must have evaluable or measurable disease according to the revised IWG Response Criteria for Malignant Lymphoma[38]. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
3. CD22 expression

   •Subjects with ALL: CD22 positive expression on malignant cells is required and must be detected by immunohistochemistry or flow cytometry. The choice of whether to use flow cytometry or immunohistochemistry will be determined by what is the most easily available tissue sample in each subject.

   CD22 expression must be demonstrated subsequent to any anti-CD22 targeted therapy (e.g. Moxetumomab pasudotox or inotuzumab ogozamicin) in subjects with ALL.

   •Subjects with aggressive B-cell NHL: CD22 expression at any level, including undetectable, will be acceptable. Subjects must have archival tissue available for analysis of CD22 expression or must be willing to undergo a biopsy of easily accessible disease.
4. Prior Bone Marrow-Stem Cell Transplant Subjects who have undergone autologous SCT with disease progression or relapse following SCT are eligible. Subjects who have undergone allogeneic SCT will be eligible if, in addition to meeting other eligibility criteria, they have no evidence of GVHD and have been without immunosuppressive agents for at least 30 days.
5. Prior Therapy Wash-out At least 2 weeks or 5 half lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy, which requires 5 half lives.

   Exceptions:
   1. There is no time restriction with regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects of such;
   2. Subjects receiving hydroxyurea may be enrolled provided there has been no increase in dose for at least 2 weeks prior to starting apheresis;
   3. Subjects who are on standard ALL maintenance type chemotherapy (vincristine, 6-mercaptopurine or oral methotrexate) may be enrolled provided that chemotherapy is discontinued at least 1 week or 5 half lives, whichever is shorter, prior to apheresis.
   4. Subjects receiving steroid therapy at physiologic replacement doses only are allowed provided there has been no increase in dose for at least 2 weeks prior to starting apheresis;
   5. For radiation therapy: Radiation therapy must have been completed at least 3 weeks prior to apheresis, with the exception that there is no time restriction if the volume of bone marrow treated is less than 10% and also the subject has measurable/evaluable disease outside the radiation port or the site of radiation has documented progression.
6. Prior CAR Therapy Subjects who have undergone prior CAR therapy must be at least 30 day post CAR infusion and have < 5% of CD3+ cells express the previous CAR if a validated assay is available.
7. Toxicities due to prior therapy must be stable or resolved (except for clinically non significant toxicities such as alopecia or cytopenias covered in *footnote to #10)
8. Age greater than or equal to 18 years of age
9. Eastern cooperative oncology group (ECOG) performance status of 0, 1, or 2; or Karnofsky ≥ 60% (See section 13.1, Appendix A)
10. Normal Organ and Marrow Function (supportive care is allowed per institutional standards, i.e. filgrastim, transfusion)

    * ANC ≥ 750/uL*
    * Platelet count ≥ 50,000/uL*
    * Absolute lymphocyte count (ALC) ≥ 150/uL*

    Adequate renal, hepatic, pulmonary and cardiac function defined as:
    * Creatinine ≤ 2 mg/dL OR creatinine clearance ≥ 60 mL/min
    * Serum ALT/AST ≤ 10x Upper limit of normal (ULN) (Elevated ALT/AST related to leukemia involvement of the liver will not disqualify a subject).
    * Total bilirubin ≤ 1.5 mg/dL, except in subjects with Gilbert's syndrome.
    * Cardiac ejection fraction ≥ 45%, no evidence of physiologically significant pericardial effusion as determined by an ECHO, MUGA or Cardiac MRI [performed within 180 days or after most recent anthracycline based treatment or mediastinal radiation therapy (whichever is most recent)]
    * No clinically significant ECG findings
    * No clinically significant pleural effusion
    * Baseline O2 saturation > 92% on room air * ALL subjects will not be excluded because of pancytopenia ≥ Grade 3 if it is felt by the investigator to be due to underlying leukemia.
11. CNS Status Subjects with CNS involvement are eligible as long as there are no overt signs or symptoms that in the evaluation of the investigator would mask or interfere with the neurological assessment of toxicity.
12. Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to leukapheresis(females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
13. Contraception Subjects of child bearing or child fathering potential must be willing to practice birth control from the time of enrollment on this study and for four (4) months after receiving the preparative lymphodepletion regimen.
14. Ability to give informed consent. Must be able to give informed consent. Legal authorized representative (LAR) is permitted if subject is cognitively able to provide verbal assent.

Exclusion criteria.

1. Recurrent or refractory ALL limited to isolated testicular disease.
2. Hyperleukocytosis (≥ 50,000 blasts/μL) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy.
3. History of other malignancy, unless disease free for at least 3 years. At the discretion of the Principal Investigator, subjects in remission for 1-2 years prior to enrollment may be deemed eligible after considering the nature of other malignancy, likelihood of recurrence during one year following CAR therapy, and impact of prior treatment on risk of CD22-CAR T cells. Subjects in remission <1 year are not eligible.

   * Exception: Nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) is eligible.
   * Hormonal therapy in subjects in remission > 1 year will be allowed.
4. Presence of active fungal, bacterial, viral, or other infection requiring intravenous antimicrobials. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
5. No knowledge of:

   * HIV,
   * Hepatitis B (HBsAg positive) or
   * Hepatitis C virus (anti HCV positive) infection. A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
6. Presence of cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement that in the judgment of the investigator may impair the ability to evaluate neurotoxicity.
7. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
8. Any medical condition that in the judgement of the sponsor investigator is likely to interfere with assessment of safety or efficacy of study treatment.
9. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
10. Women who are pregnant or breastfeeding.
11. In the investigator's judgment, the subject is unlikely to complete all protocol required study visits or procedures, including follow up visits, or comply with the study requirements for participation.
12. Primary immunodeficiency or history of autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Rate of successful manufacture of CD22 CAR T cells | 7-11 days from start of manufacturing
  The percentage of apheresis samples (fresh or frozen) that are successfully processed and expanded to manufacture CD22 CAR T cells will be determined for each dose cohort.
MTD/RP2D of CD22-CAR T cells in subjects with aggressive B-cell NHL | 28 days after infusion of CD22 CAR T cells
  Incidence and severity of dose limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD22 CAR T cells, as recorded and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, at each dose level tested in subjects with aggressive B-cell NHL
Safety evaluation of CD22-CAR T cells in subjects with ALL | 2 years after infusion of CD22-CAR T cells
  Incidence and severity of dose limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD22 CAR T cells, as recorded and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, at each dose level tested in subjects with ALL

SECONDARY OUTCOMES:
Clinical activity of CD22-CAR T cells in adults with relapsed/refractory CD22-expressing B-cell ALL at target dose | 28 months after infusion of CD22-CAR T cells
  Clinical activity will be assessed by modified International Working Group response criteria for acute lymphoblastic leukemia. Results will be reported as best response (i.e. complete response (CR), partial response (PR), stable disease )SD), or progressive disease [PR]) at Day 28 for adult subjects with ALL treated at the target dose.
Clinical activity of CD22-CAR T cells in adults with relapsed/refractory aggressive B-cell NHL at MTD/RP2D | 3 months after infusion of CD22-CAR T cells
  Clinical activity will be assessed by Lugano response criteria for lymphoma (see Appendix 13.3.2). Results will be reported as best response (i.e. complete response [CR], partial response [PR], stable disease [SD], or progressive disease [PR]) at Month 3 for adult aggressive B-cell NHL subjects treated at MTD/RP2D.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Frank, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frank MJ, Baird JH, Kramer AM, Srinagesh HK, Patel S, Brown AK, Oak JS, Younes SF, Natkunam Y, Hamilton MP, Su YJ, Agarwal N, Chinnasamy H, Egeler E, Mavroukakis S, Feldman SA, Sahaf B, Mackall CL, Muffly L, Miklos DB; CARdinal-22 Investigator group. CD22-directed CAR T-cell therapy for large B-cell lymphomas progressing after CD19-directed CAR T-cell therapy: a dose-finding phase 1 study. Lancet. 2024 Jul 27;404(10450):353-363. doi: 10.1016/S0140-6736(24)00746-3. Epub 2024 Jul 9. PMID 38996463
- [Derived] Baird JH, Frank MJ, Craig J, Patel S, Spiegel JY, Sahaf B, Oak JS, Younes SF, Ozawa MG, Yang E, Natkunam Y, Tamaresis J, Ehlinger Z, Reynolds WD, Arai S, Johnston L, Lowsky R, Meyer E, Negrin RS, Rezvani AR, Shiraz P, Sidana S, Weng WK, Davis KL, Ramakrishna S, Schultz L, Mullins C, Jacob A, Kirsch I, Feldman SA, Mackall CL, Miklos DB, Muffly L. CD22-directed CAR T-cell therapy induces complete remissions in CD19-directed CAR-refractory large B-cell lymphoma. Blood. 2021 Apr 29;137(17):2321-2325. doi: 10.1182/blood.2020009432. PMID 33512414